CLINICAL TRIAL: NCT03950544
Title: How to Optimize the Combined Antibiotic Therapy for Carbapenem Resistant Klebsiella Pneumoniae
Brief Title: The Combined Antibiotic Therapy for Carbapenem Resistant Klebsiella Pneumoniae
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sheng Wang MD PhD, Director, Shanghai 10th People's Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STPH-ICU-002
Record Dates: First submitted 2018-10-30; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Antibiotic Resistant Infection
MeSH Terms: interventions — Fosfomycin; Meropenem; Tigecycline; Polymyxin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- only meropenem therapy, (Experimental): this group is only meropenem therapy as a single antibiotic treatment
  Interventions: Drug: Fosfomycin; Drug: Tigecycline; Drug: Polymyxin B

INTERVENTIONS:
Drug: Fosfomycin — Fosfomycin and meropenem
  Other Names: meropenem
Drug: Tigecycline — Tigecycline and meropenem
  Other Names: meropenem
Drug: Polymyxin B — Polymyxin B and meropenem
  Other Names: meropenem

SUMMARY:
The infection of carbapenem resistant klebsiella pneumoniae (CRKP) is increasingly serious.Based on the early experimental basis and relevant research background,this study intends to separate and purify the CRKP from the bronchoalveolar lavage fluid (BALF) of the clinical patients.Designed by checkerboard assay and time-kill assay(TKA)，this study can explore the best combination therapy based on carbapenems.

DETAILED DESCRIPTION:
1. Collect the BALF from patients diagnosed with CRKP infection in surgical intensive care unit（SICU）of Shanghai 10th people's hospital.
2. Separate and purify the BALF. Divide each CRKP into four treatment groups based on meropenem.

3.1 By checkerboard method and microdilution broth method,get the minimal inhibitory concentration (MICS) of two antibiotics,then calculate the fractional inhibitory concentration (FIC) index according to MIC results.

3.2 Observe the effect of two antibiotics on the growth of CRKP by TKA.

4.By the above two invitro experiments, analyze the data of the experimental results and get the best combination therapy based on carbapenems.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 90.
* infected with CRKP firstly .

Exclusion Criteria:

* APACHE II score > 35
* Vital signs are unstable
* Unable to tolerate fiberoptic bronchoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the fractional inhibitory concentration index (FICI) | 24hours-36hours
  By checkerboard method and microdilution broth method,get the minimal inhibitory concentration (MICS) of two antibiotics,then calculate the fractional inhibitory concentration (FIC) index according to MIC results.
  Evaluation index:
  FIC=0.5 , coordinating effect. 0.5 < FIC <1, adding effect;
  1 < FIC <2, irrelevant.

SECONDARY OUTCOMES:
the time-kill assay (TKA) | 36hours-48hours
  According to the Clinical and Laboratory Standards Institute,observe the changes of bacterial growth over time after different combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Li Hua, master, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du Y, Mu S, Liu Y, Yuan Y, Zhu Y, Ma L, Wang Q, Zhu Z, Liu Y, Wang S. The Genomic Characterization of KPC-Producing Klebsiella pneumoniae from the ICU of a Teaching Hospital in Shanghai, China. Infect Drug Resist. 2022 Jan 11;15:69-81. doi: 10.2147/IDR.S343673. eCollection 2022. PMID 35046672